CLINICAL TRIAL: NCT03242785
Title: Impact of Self-monitoring of Blood Pressure and Self-titration of Antihypertensive Medication in the Control of Hypertension and Adherence to Treatment. A Pragmatic, Randomized, Controlled Clinical Trial (ADAMPA Study).
Brief Title: Impact of Self-monitoring of Blood Pressure and Self-titration of Medication in the Control of Hypertension (ADAMPA)
Acronym: ADAMPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, José Sanfelix, Primary Care Physician, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ADAMPA; 2016-003986-25 (EudraCT Number)
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Hypertension; Adjustment; Adherence, Medication
Keywords: Self-monitoring; Education; Self-titration; antihypertensives
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-monitoring/Self-titration (Experimental): The intervention consists of self-monitoring blood pressure at home, and subsequent medication self-titration, based on a medication adjustment plan pre-established by the family physician, in patients with uncontrolled hypertension.
  Interventions: Other: Self-monitoring/Self-titration
- Routine care (No Intervention): Patients in this arm will receive routine care for high blood pressure in the primary health care center.

INTERVENTIONS:
Other: Self-monitoring/Self-titration — The intervention of the ADAMPA trial is not pharmacological but an intervention that modifies usual clinical practice. The intervention of self-monitoring and self-titration of the medication is composed of 3 elements:
  1. Education of the patient: information and training on hypertension, its risks, management, the benefits of an adequate control and the generic measures for an optimal control.
  2. Training for self-monitoring: Patients will be trained to perform the self-measurement of blood pressure correctly (and recording their values in the sheet enabled for this purpose)
  3. Training for self-titration: patients will be instructed on the target BP numbers, individualized for each patient, on the mode of action against specific figures, including self-adjustment of drug treatment.
  Arms: Self-monitoring/Self-titration

SUMMARY:
The ADAMPA study is a pragmatic randomized clinical trial which aims to evaluate the effectiveness of an intervention based on self-monitoring and self-titration of medication in poorly controlled hypertensive patients 40 years and older. The total duration of the study is 3 years, with 6 months of enrolment and 1 year of follow-up to measure the primary endpoint (Difference in mean systolic blood pressure, in mmHg, between the intervention and control groups).

DETAILED DESCRIPTION:
ADAMPA study. Objectives: To evaluate the comparative effectiveness of an intervention that includes educational components, self-monitoring of blood pressure and self-titration of antihypertensive medication in the improvement of control of hypertension compared to usual care in a poorly controlled population of hypertensive patients.

Design: Pragmatic, controlled, randomized, non-masked clinical trial with two parallel arms.

Disease related to the study: Hypertension.

Main outcome measure: Difference in mean systolic blood pressure, in mmHg. At 12 months of follow-up between the intervention and control groups, determined at physicians' practice with a validated automatic electronic sphygmomanometer

Study population: Patients assigned to the Valencia Clinic-La Malvarrosa Health Department. Total number of patients to be randomized: 458 (229 per arm).

Duration of intervention: 12 months (also, a pragmatic extension with passive follow-up is planned for 24 months, collecting a reduced set of outcome variables, as secondary variables)

Calendar and expected completion date: The trial will take place over 3 years (6 months of recruitment, 12 months of follow-up for the main analysis of results, 12 months of pragmatic follow-up at 24 months, and finally 6 months for reporting results). Estimated Completion Date: 2020.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older
* Diagnosis of hypertension of any origin
* Systolic blood pressure (SBP) > 145 or diastolic blood pressure (DBP) > 90 mm Hg at baseline
* Voluntarily participation in the study and having signed the corresponding informed consent.

Exclusion Criteria:

* Inability to understand and/or perform self-adjustment of the medication, including dementia or significant cognitive impairment (at the discretion of the investigator performing the recruitment).
* History of orthostatic hypotension (fall> 20 mm Hg in SBP after adopting the orthostatic position).
* SBP> 200 or DBP> 100 mm Hg on the baseline examination
* Being on treatment with more than 4 antihypertensive drugs
* Participation in another study on high blood pressure or in a clinical trial
* Presence of tremor or neurological disease that makes it difficult to perform BP self-measurement.
* Presence of arrhythmia
* Presence of terminal illness
* Chronic disability impeding to leave home
* History of acute cardiovascular event in the last 3 months
* Hypertension managed directly by specialist physicians outside the primary care setting.
* Spouse selected for the study
* Non-resident or transient patients
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure (SBP). | 12 months from start of intervention
  Difference in mean systolic blood pressure, in mmHg. At 12 months of follow-up between the intervention and control groups, determined at physicians' practice with a validated automatic electronic sphygmomanometer

SECONDARY OUTCOMES:
Mean systolic blood pressure at 6 and 24 months | 6 and 24 months
  Difference in mean systolic blood pressure, in mmHg at 6 and 24 months of follow-up between intervention and control groups determined at physicians' practice with a validated automatic electronic sphygmomanometer
Mean diastolic blood pressure (DBP) at 6 and 24 months | 6 and 24 months
  Difference in mean diastolic blood pressure, in mmHg at 6 and 24 months of follow-up between intervention and control groups determined at physicians' practice with a validated automatic electronic sphygmomanometer
Percentage of patients with normal SBP and DBP | 6,12, 24 months
  Percentage of patients with SBP<140 mmHg and DBP <90 mmHg at 6, 12 y 24 months of follow-up
EuroQoL-5D score | 6,12,24 months
  Score in the EuroQoL-5D at 6, 12 and 24 months of follow-up
Medication adherence | 12 months
  Proportion of days covered (PDC) will be measured, dividing the number of days with dispensed medication by the number of days of follow-up. Patients with PDC ≥ 80 will be considered adherent. In case of polypharmacy, patients with PDC ≥ 80 for all the medications will be considered adherent.
Medication persistence | 12 months
  Persistence will be defined as the time of continuous utilization of the correspondent medication from the start of follow-up until its discontinuation (when the patient stops picking up the medication after a 60-days grace period, once the period with available medication from the previous dispensation is finished).
Therapeutic inertia | 6,12,24 months
  Defined as the quotient resulting of dividing the number of patients whose pharmacological treatment has not been modified, by the number of patients with SBP and/or DBP measured in the physician's practice, with values above the recommendations of the European Society of Hypertension and European Society of Cardiology. This measurements will be performed at 6, 12 and 24 months.

OTHER OUTCOMES:
Changes in lifestyle | 6,12,24 months
  Changes in lifestyle (smoking, exercise, body weight) at 6, 12, and 24 months compared to these characteristics at baseline.
Adverse events | 12 months
  We will assess if any of the following adverse events are present during the follow-up: angor, myocardial infarction, stroke, hypotensive crisis and death.
Health services utilization | 6,12 and 24 months
  Health services utilization during follow-up (6, 12 and 24 months), will include: visits to primary care nurse and physician, related to high blood pressure (HBP) (including telephone and home), emergency visits to hospital, hospital admissions, hospitalization days per admission and principal diagnosis.
Incremental cost per quality-adjusted life year gained | 12 months
  Incremental cost per quality-adjusted life year gained in the intervention group as compared to the control group.
Satisfaction with the intervention | 12 months
  Qualitative evaluation of the intervention by patients and research physicians, through a satisfaction scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sanfélix-Gimeno, Dr, Principal Investigator — Health Services Research Unit FISABIO
Locations (1):
- Departamento de Salud Valencia Clínico Malvarrosa, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Ibanez P, Marco-Moreno I, Garcia-Sempere A, Peiro S, Martinez-Ibanez L, Barreira-Franch I, Bellot-Pujalte L, Avelino-Hidalgo E, Escrig-Veses M, Boveda-Garcia M, Calleja-Del-Ser M, Robles-Cabaninas C, Hurtado I, Rodriguez-Bernal CL, Gimenez-Loreiro M, Sanfelix-Gimeno G, Sanfelix-Genoves J; ADAMPA Research Group. Long-Term Effect of Home Blood Pressure Self-Monitoring Plus Medication Self-Titration for Patients With Hypertension: A Secondary Analysis of the ADAMPA Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2410063. doi: 10.1001/jamanetworkopen.2024.10063. PMID 38728033
- [Derived] Martinez-Ibanez P, Marco-Moreno I, Peiro S, Martinez-Ibanez L, Barreira-Franch I, Bellot-Pujalte L, Avelino-Hidalgo E, Escrig-Veses M, Boveda-Garcia M, Calleja-Del-Ser M, Ferrero-Gregori A, Iftimi AA, Hurtado I, Garcia-Sempere A, Rodriguez-Bernal CL, Gimenez-Loreiro M, Sanfelix-Gimeno G, Sanfelix-Genoves J; ADAMPA research group. Home Blood Pressure Self-monitoring plus Self-titration of Antihypertensive Medication for Poorly Controlled Hypertension in Primary Care: the ADAMPA Randomized Clinical Trial. J Gen Intern Med. 2023 Jan;38(1):81-89. doi: 10.1007/s11606-022-07791-z. Epub 2022 Oct 11. PMID 36219303